CLINICAL TRIAL: NCT06944223
Title: Oxalate and Citrate in Humans - Response to Citrate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB25-0030; 5K23DK127252-03 (NIH)
Record Dates: First submitted 2025-04-17; First posted 2025-04-25 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Kidney Stone; Healthy
Keywords: kidney stone; kidney stones
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kidney stone formers (Other): 12 stone-forming subjects will be enrolled in this arm.
  Interventions: Other: Kidney stone formers
- Control cohort (Other): 12 non-stone-forming subjects will be enrolled in this arm.
  Interventions: Other: Control cohort

INTERVENTIONS:
Other: Kidney stone formers — Consuming a special drink (potassium citrate) during an all-day visit to the University of Chicago research clinic
  Subjects in both groups will be asked to partake in the same activities, as follows: The day before presenting to the research clinic, subjects will collect urine at home. Subjects will then come to the research clinic at the University of Chicago in Hyde Park, where they will spend most of the day. We will give them a special liquid that contains potassium citrate. After this, we will collect urine and blood samples throughout the day. While at the clinic, subjects will also receive a boxed lunch at the end of the visit.
  Arms: Kidney stone formers
Other: Control cohort — Consuming a special drink (potassium citrate) during an all-day visit to the University of Chicago research clinic
  Subjects in both groups will be asked to partake in the same activities, as follows: The day before presenting to the research clinic, subjects will collect urine at home. Subjects will then come to the research clinic at the University of Chicago in Hyde Park, where they will spend most of the day. We will give them a special liquid that contains potassium citrate. After this, we will collect urine and blood samples throughout the day. While at the clinic, subjects will also receive a boxed lunch at the end of the visit.
  Arms: Control cohort

SUMMARY:
This is a single-center study that aims to learn more about how two compounds found in food, oxalate and citrate, interact in the body and may influence a person's chances of forming kidney stones. The study will examine changes in urinary oxalate and citrate levels after participants consume potassium citrate.

DETAILED DESCRIPTION:
Administration of oral potassium citrate without oxalate is the next step in determining whether there is a transporter-mediated mechanism linking urinary oxalate and citrate excretion in humans. The study investigators will measure the fractional excretion (FE) of oxalate and citrate. Both substances are freely filtered by the renal glomerulus and are subsequently either secreted or reabsorbed (oxalate), or reabsorbed (citrate). By calculating fractional excretion, the investigators will assess urinary excretion relative to filtered load and tubular handling.

Experimental Design:

Studies will be conducted at the University of Chicago Medicine (UCM) Clinical Research Center (CRC).

Informed Consent Process:

Participants will undergo the informed consent process with either the principal investigator or the study research assistant. Participants will be given ample time to ask questions and discuss the study. No research activities will occur before the consent form is signed.

In participants with no history of kidney stones (non-stone formers [NSF], N=12) and participants with a history of calcium oxalate kidney stones (CaOx stone formers [SF], N=12), the investigators will administer a single dose of oral potassium citrate and measure both urine and blood levels of oxalate and citrate over six hours.

Primary endpoint (Hypothesis 1a): Change from baseline in fractional excretion of oxalate, adjusted for change in fractional excretion of citrate, following the potassium citrate load.

Secondary endpoint (Hypothesis 1b): Comparison of the adjusted change in fractional excretion of oxalate in calcium stone formers versus non-stone formers.

Rationale:

There is a known association between urinary oxalate and citrate excretion. A prior study conducted by the research team involved administering an oral oxalate load to calcium stone formers and non-stone formers. The results showed a correlated increase in urinary citrate excretion following the oxalate load. If this is due to specific effects of oxalate and citrate transporters in the proximal renal tubule, then administering a potassium citrate load should increase urinary oxalate excretion. Furthermore, this increase may differ between non-stone formers and stone formers.

Hypothesis 1a: An oral potassium citrate load will increase fractional excretion of oxalate.

Hypothesis 1b: The increase will be greater in non-stone formers than in calcium oxalate stone formers who are non-obese.

If these hypotheses are correct, this would suggest a role for proximal tubule transporter proteins-specifically solute carrier family 26 member 6 (SLC26A6) and sodium-dependent dicarboxylate cotransporter 1 (NaDC1)-in coordinating oxalate and citrate handling. If not, other factors such as dietary differences may explain the association.

Study Population and Recruitment:

A total of 24 participants will be enrolled (12 non-stone formers, 12 stone formers), balanced by sex, over the first two years of the study award period.

Non-stone formers will be recruited from a pool of previous research participants, as well as via ResearchMatch and The New Normal, two UCM Institute for Translational Medicine resources used to connect researchers with individuals interested in research participation. These platforms will be queried to identify eligible controls.

Eligible non-stone former controls must complete a home 24-hour urine collection to screen for abnormal acid-base balance or oxalate excretion.

Stone formers, all of whom will have existing 24-hour urine data, will be recruited from the UCM Kidney Stone Clinic (both current patients and the repository of past patients). This clinic has maintained patient records for over 50 years and is a reliable source of research participants for this study group.

Inclusion Criteria:

Stone formers (SF): Age 18-70; history of at least one calcium-based kidney stone.

Non-stone formers (NSF): Age 18-70; no history of kidney stones; 24-hour urinary oxalate within laboratory reference range (<50 mg/day).

Exclusion Criteria:

History of primarily uric acid, cystine, or struvite kidney stones.

History of severe acid-base abnormalities.

24-hour urinary citrate <100 mg/day or >1500 mg/day.

Use of diuretic medications or alkali supplements that cannot be safely discontinued for the study period.

Chronic kidney disease (glomerular filtration rate <75 mL/min/1.73 m²).

NSF or SF participants with extreme urinary citrate values will be excluded to minimize variability and focus on typical ranges.

Protocol:

This protocol builds on previously published studies and an Institutional Review Board (IRB)-approved study (IRB# 21-1349) that involved administering an oxalate load to similar populations. Stone formers both on and off alkali therapy will be included. Those on alkali therapy will be asked to discontinue their supplement for two weeks prior to the study day. All participants will be asked to hold vitamin C, multivitamins, calcium supplements, and diuretics for one week prior to the study. Medication adjustments will be made in consultation with each participant's primary care physician or nephrologist.

One day before the study visit, participants will complete a home 24-hour urine collection and a food frequency questionnaire. On the study day, participants will be admitted to the UCM Clinical Research Center in a fasting state. Three baseline urine and blood samples will be collected, and height and weight will be recorded. Participants will then ingest 40 milliequivalents (mEq) of oral potassium citrate.

Urine and blood will be collected every 45 minutes for six hours following the dose. Each blood draw will require approximately 8 mL of blood (total of 9 draws). Participants will remain fasting throughout the study. They will be provided with 500 mL of water at the start, and may drink additional water as desired. A boxed lunch will be offered at the end of the study.

Urine and Serum Measurements:

24-hour and timed urine samples will be collected and analyzed for oxalate and citrate, along with other stone risk factors: urine volume, calcium, pH, uric acid, sodium, potassium, chloride, magnesium, phosphorus, urea, sulfate, ammonium, and creatinine.

Supersaturation of calcium oxalate, calcium phosphate, and uric acid will be calculated using the EQUIL2 program.

Serum measurements will include sodium, potassium, chloride, bicarbonate, calcium, phosphorus, magnesium, creatinine, as well as oxalate and citrate.

Urine and serum samples will be processed at the UCM Kidney Stone Laboratory, except for plasma oxalate, which will be analyzed at the University of Alabama at Birmingham (UAB). Samples will be stored at -80°C for potential future use.

Clinical Variable Collection:

Demographic and clinical variables-including age, sex, height, weight, body mass index (BMI), chronic medical conditions, and medications-will be extracted from the electronic medical record and verified via participant interview.

Statistical Analysis:

Changes from baseline in urinary oxalate, urinary citrate, and fractional excretion of both analytes will be calculated for each time point. Descriptive statistics and t-tests will be used to assess changes in excretion patterns within and between stone formers and non-stone formers. Graphs will depict the time-course of these changes. Longitudinal regression models will assess associations between urinary oxalate and citrate excretion, stratified by stone-forming status. Multivariate analyses will include clinical (e.g., sex, BMI) and urinary variables (e.g., gastrointestinal anion excretion).

Sample Size and Power Calculation:

Sample size was determined using preliminary data demonstrating a between-group difference in the ratio of change in citrate (millimoles)/creatinine to change in oxalate (millimoles)/creatinine. In non-stone formers, this ratio was 3.0 (standard deviation 1.5), compared to 0.3 (standard deviation 0.1) in stone formers. Assuming an alpha of 0.05 and 80% power, 12 participants per group (total N=24) will provide sufficient power to detect this difference.

ELIGIBILITY:
Inclusion Criteria:

Stone formers (SF):

* Age 18-70
* History of at least one calcium-based kidney stone

Non-stone formers (NSF):

* Age 18-70
* No history of kidney stone
* 24-hour urine oxalate within laboratory normal range (<50 mg/day)

Exclusion Criteria:

History of primarily uric acid, cysteine, or struvite stones

History of severe acid-base abnormality, very low (less than 100 mg/day) or very high (greater than 1500 mg/day) urine citrate

Any controls or stone former (SF) participants who cannot stop diuretic medication or alkali supplementation for the course of the study period

Chronic kidney disease (glomerular filtration rate <75 milliliters per minute per 1.73 square meters [mL/min/1.73 m²])

Non-stone formers (NSF) and stone formers (SF) with extreme levels of urine citrate will be excluded from this small initial study to reduce heterogeneity and remove focus from the extremes of citrate levels.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in urine oxalate from baseline to 2-hours, 4-hours, and 6-hours after potassium citrate consumption. | 6 hours
  Urine oxalate will be measured or calculated at time points 0, 2-hours, 4-hours, and 6-hours after sodium oxalate consumption. We will compare change in urine citrate and fractional excretion of citrate by change in oxalate at each time period for all participants.
Change in urine citrate from baseline to 2-hours, 4-hours, and 6-hours after potassium citrate consumption. | 6 hours
  Urine citrate will be measured or calculated at time points 0, 2-hours, 4-hours, and 6-hours after sodium oxalate consumption. We will compare change in urine citrate and fractional excretion of citrate by change in oxalate at each time period for all participants.
Change in fractional excretions of citrate and oxalate from baseline to 2-hours, 4-hours, and 6-hours after potassium citrate consumption. | 6 hours
  Fractional excretion of citrate will be measured or calculated at time points 0, 2-hours, 4-hours, and 6-hours after sodium oxalate consumption. We will compare change in urine citrate and fractional excretion of citrate by change in oxalate at each time period for all participants.

SECONDARY OUTCOMES:
Difference in change in urine oxalate from baseline between kidney stone patients and controls. | 6 hours
  We will compare change urine citrate and fractional excretion of citrate by change in oxalate at each time period (0 to 2-hours, 4-hours, and 6-hours) between kidney stone patients and controls
Difference in change in urine citrate from baseline between kidney stone patients and controls. | 6 hours
  We will compare change urine citrate and fractional excretion of citrate by change in oxalate at each time period (0 to 2-hours, 4-hours, and 6-hours) between kidney stone patients and controls.
Difference in change in fractional excretions of citrate and oxalate from baseline between kidney stone patients and controls. | 6 hours
  We will compare change urine citrate and fractional excretion of citrate by change in oxalate at each time period (0 to 2-hours, 4-hours, and 6-hours) between kidney stone patients and controls.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States